CLINICAL TRIAL: NCT03238664
Title: Robot-Assisted Laparoscopic HIFU (High-Intensity Focused Ultrasound) of the Bladder Wall for Thermal Ablation of Muscle Invasive Cells of Bladder Tumors: Corroborating With Robot-Assisted Radical Cystectomy
Brief Title: Robot-Assisted Laparoscopic High-Intensity Focused Ultrasound and Radical Cystectomy for Thermal Ablation of Muscle Invasive Cells in Patients With Bladder Tumors
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No funding
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4B-15-6; NCI-2017-00626 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 4B-15-6 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2017-07-31; First posted 2017-08-03 (Actual); Last update posted 2018-01-02 (Actual); Status verified 2017-12

CONDITIONS: Infiltrating Bladder Urothelial Carcinoma; Stage II Bladder Urothelial Carcinoma; Transitional Cell Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — Biopsy; High-Intensity Focused Ultrasound Ablation; Extracorporeal Shockwave Therapy; Cystectomy; Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Arm A (laparoscopic HIFU, RARC) (Experimental): Patients undergo pre-HIFU CEUS, standard of care biopsy of the bladder tumor, laparoscopic HIFU, and post-HIFU CEUS. Patients then undergo standard of care RARC.
  Interventions: Procedure: Biopsy; Device: High-Intensity Focused Ultrasound Ablation; Other: Laboratory Biomarker Analysis; Procedure: Radical Cystectomy; Device: Ultrasonography
- Arm B (RARC) (Active Comparator): Patients undergo standard of care RARC.
  Interventions: Other: Laboratory Biomarker Analysis; Procedure: Radical Cystectomy

INTERVENTIONS:
Procedure: Biopsy — Undergo biopsy of bladder tumor
  Other Names: Bx
  Arms: Arm A (laparoscopic HIFU, RARC)
Device: High-Intensity Focused Ultrasound Ablation — Undergo laparoscopic HIFU
  Other Names: HIFU; high-intensity focused ultrasound therapy
  Arms: Arm A (laparoscopic HIFU, RARC)
Other: Laboratory Biomarker Analysis — Correlative studies
Procedure: Radical Cystectomy — Undergo RARC
  Other Names: Complete Cystectomy
Device: Ultrasonography — Undergo CEUS
  Other Names: 2-Dimensional Grayscale Ultrasound Imaging; 2-Dimensional Ultrasound Imaging; 2D-US; Ultrasound; Ultrasound Imaging; Ultrasound Test; Ultrasound, Medical; US
  Arms: Arm A (laparoscopic HIFU, RARC)

SUMMARY:
This randomized pilot trial studies how well robot-assisted laparoscopic high-intensity focused ultrasound works compared to robot-assisted radical cystectomy for thermal ablation of muscle invasive cells in patients with bladder tumors. Laparoscopic high-intensity focused ultrasound uses high frequency sound waves to deliver a strong beam to a specific part of the tumor and may lower the number of tumor cells released into the blood stream compared to radical cystectomy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To obtain preliminary estimates of the efficacy of laparoscopic high-intensity focused ultrasound (HIFU) for the treatment of localized primary bladder cancer.

II. To estimate the change in the number of expelled circulating tumor cells (CTCs), when comparing HIFU to robot-assisted radical cystectomy (RARC) alone.

SECONDARY OBJECTIVES:

I. To evaluate the safety and toxicity of using laparoscopic HIFU.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo pre-HIFU contrast-enhanced ultrasound (CEUS), standard of care biopsy of the bladder tumor, laparoscopic HIFU, and post-HIFU CEUS. Patients then undergo standard of care RARC.

ARM B: Patients undergo standard of care RARC.

After completion of study, patients are followed up at 2 weeks and 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Must meet all inclusion and exclusion criteria
* Presence of a muscle invasive bladder tumor(s) (T2), specific for transitional cell carcinoma on pre-operative histology (i.e. biopsy or transurethral resection of bladder tumor [TURBT]).
* Presence of a single bladder tumor lesion
* Patients are scheduled to undergo RARC at our institution
* Subjects must have given written informed consent to agree to participate
* Previous chemotherapy, and/or biological therapy for cancer are permitted provided that the acoustic properties of the tumor were not affected, but the subject should have recovered from the effects of these or of any prior surgery; chemotherapy can be within 70 days of operation
* Subjects must be free of any clinically significant disease other than cancer that would interfere with the study evaluations
* Pre-operative computed tomography (CT)/magnetic resonance imaging (MRI) abdomen and pelvis within 90 days
* Absolute neutrophil count (ANC) >= 1500 mm^-3
* Platelet count >= 100,000 mm^-3
* Hemoglobin >= 10 g/dl
* Prothrombin time (PT) =< 1.5 times upper limit of laboratory normal (ULN)
* Activated partial thromboplastin time =< 1.5 times ULN
* Total bilirubin < 1.5 times ULN
* Aspartate aminotransferase (AST) =< 3 times ULN
* Alkaline phosphatase < 2 times ULN, unless arising from bone

Exclusion Criteria:

* Subjects deemed unsuitable candidates and not medically optimized for RARC
* Subjects with tumors lying < 1 cm from sensitive structures such as the ureter, prostate or adjacent bowel
* Patients with presence of multiple bladder lesions
* Subjects on concurrent anticoagulant, or immunosuppressive medication
* Patients with pre-operative histologic confirmation of a bladder lesion other than transitional cell carcinoma
* Subjects on anti-cancer medication whether biologic or pharmaceutical
* Women who are pregnant or nursing (pregnancy test to be performed within 24 hours prior to HIFU treatment)
* Subjects assessed by consultant anesthetist as unsuitable for general anesthetic
* Absolute contraindications: venous injury at the level of the femoral veins or proximally; known or suspected thrombosis of the femoral or iliac veins on the proposed side of venous cannulation, ambulatory patient
* Relative contraindications: presence of bleeding disorders; distortion of anatomy due to local injury or deformity; previous long-term venous catheterization; history of vasculitis; previous injection of sclerosis agents; previous radiation therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-01-22 (Estimated); Primary Completion 2019-01-22 (Estimated); Study Completion 2020-01-22 (Estimated)

PRIMARY OUTCOMES:
Complete ablation of the targeted lesion in the bladder wall assessed by histopathologic examination and Live/Dead Viability/Cytotoxicity Assay Kit of the resected specimen (Arm A) | At the day of surgery
  A Clopper-Pearson (exact) 90% confidence interval will be constructed for the probability of a successful HIFU procedure.
CTC enumeration assessed using quantitative real-time polymerase chain reaction | Up to 7 days post-surgery
  The mean number of CTCs in each patient, as well as the difference between the two arms (possibly after log or square root transformation) will be estimated. Importantly the numbers of CTCs captured in the femoral lines will be compared to the numbers captured in the peripheral lines. Means and 90% confidence intervals will be calculated. Changes in CTC enumeration in a group that undergoes HIFU (Arm A) to a group that does not undergo HIFU (Arm B) will be observed.

SECONDARY OUTCOMES:
Incidence of adverse events evaluated according to National Cancer Institute Criteria for Adverse Events version 4.0 (Arm A) | Up to 3 months
  The complication observed in all patents in each arm will be reported and summarized. For Arm A, focus will be on the complications that might be associated with the HIFU procedure; for Arm B, focus will be on the safety of placed a line in the femoral vein.

CONTACTS AND LOCATIONS:
Overall Officials: Inderbir Gill, MD, Principal Investigator — University of Southern California